CLINICAL TRIAL: NCT03443427
Title: An Observer-blind Study to Evaluate the Safety, Reactogenicity and Immunogenicity of the Investigational GSK Biologicals' COPD Vaccine (GSK3277511A) in Adults
Brief Title: A Study to Test if a Third Dose of the Vaccine is Safe in Current and Former Smokers Aged 40 to 80 Years Old and to Gather Information on the Immune Response Following the Third Dose of the Vaccine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 207759; 2017-002941-31 (EudraCT Number)
Record Dates: First submitted 2018-02-14; First posted 2018-02-23 (Actual); Results first posted 2020-11-12 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-07

CONDITIONS: Respiratory Disorders
Keywords: Non-typeable Haemophilus influenzae; Moraxella catarrhalis; Safety; Third vaccine dose; Vaccination; Immunogenicity
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: By observer-blind, it is meant that during the course of the study, the vaccine recipient and those responsible for the evaluation of any study endpoint (e.g. safety, reactogenicity) will all be unaware of whether vaccine or placebo was administered. Each study site is responsible for having a blinding plan. To work in an observer-blind manner, vaccine preparation and administration will be done by authorised medical personnel (e.g. study nurse) who will not participate in any of the study clinical evaluation assays. Two teams of study personnel will hence be set up:
  * A team of unblinded personnel (responsible for the preparation and the administration of the vaccines)
  * A team of blinded personnel (responsible for the clinical evaluation of the subjects).
  The laboratory in charge of the laboratory testing will be blinded to the treatment, and codes will be used to link the subject and study (without any link to the treatment attributed to the subject) to each sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Schedule 0-2-6 Group (Experimental): Subjects between, and including, 40 and 80 years of age at the time of the first vaccination, receiving three doses of the GSK3277511A investigational vaccine at Day 1 (Month 0), Day 61 (Month 2) and Day 181 (Month 6) and one dose of placebo at Day 361 (Month 12).
  Interventions: Biological: NTHi Mcat investigational vaccine (GSK3277511A); Biological: Placebo
- Schedule 0-2-12 Group (Experimental): Subjects between, and including, 40 and 80 years of age at the time of the first vaccination, receiving three doses of the GSK3277511A investigational vaccine at Day 1 (Month 0), Day 61 (Month 2) and Day 361 (Month 12) and one dose of placebo at Day 181 (Month 6).
  Interventions: Biological: NTHi Mcat investigational vaccine (GSK3277511A); Biological: Placebo

INTERVENTIONS:
Biological: NTHi Mcat investigational vaccine (GSK3277511A) — Two doses administered intramuscularly at Day 1 and Day 61 in the deltoid region of the non-dominant arm and a third dose administered at either Day 181 or Day 361, according to each vaccination scheduling defined per protocol.
Biological: Placebo — One dose administered intramuscularly at either Day 181 or Day 361 in the deltoid region of the non-dominant arm.

SUMMARY:
The purpose of this study is to test two different vaccine schedules to be used for administering the investigational NTHi Mcat vaccine that will be targeting patients with chronic obstructive pulmonary disease (COPD) to prevent acute exacerbations. An acute exacerbation is when the breathlessness in COPD patients will get even worse than it normally already is, sometimes to the point where oxygen therapy is required.

In previous studies, study participants have received two doses of the vaccine according to a 0, 2 month vaccination schedule, in addition to standard care. The current study will find out if a third dose of the study vaccine against NTHi/Mcat is safe and working well. The study will also investigate if the third dose of vaccine works best when given after 6 months or after 12 months.

DETAILED DESCRIPTION:
The purpose of this Phase 2 study is to evaluate two vaccine schedules of the investigational NTHi-Mcat vaccine.

As the prevalence of COPD increases with age and as age has an influence on both the immunogenicity and reactogenicity of a vaccine, subjects 40-80 years old will be enrolled. As cigarette smoking is the most commonly encountered risk factor for COPD, adults with a smoking history of at least 10 pack-years will be selected in order to immunologically match the COPD population as much as possible. Literature data indeed suggest that alterations of the immune system start early on in smokers, before the COPD disease is recognized [Barcelo et al 2008; Droemann et al, 2005; Takanashi et al, 1999].

Several formulations of a vaccine containing the NTHi antigens (10 or 30 µg) either non-adjuvanted or combined with different adjuvants (aluminium [Al], adjuvant system [AS]01E and AS04C) were already evaluated in two previous Phase 1 clinical trials (NTHI-002 in healthy adults aged 18 - 40 years and NTHI-003 in current and former healthy smokers of 50-70 years old). The investigational vaccines were well-tolerated, with an acceptable safety and reactogenicity profile. These studies allowed the dose selection of the NTHi antigens (10 µg) and the adjuvant system (AS01E) evaluated for the first time in moderate and severe COPD patients aged 40-80 years in the Phase 2 study NTHI-004.

The safety, reactogenicity and immunogenicity of different formulations of the NTHi-Mcat investigational vaccine have been evaluated in the Phase 1 study in healthy adults aged 18-40 years and in current and former smokers aged 50-70 years (study NTHI MCAT-001). Based on results obtained up to 30 days post-Dose 2 from this study, the AS01E-adjuvanted formulation containing 10 µg of NTHi proteins PD and PE-PilA and 3.3 µg of UspA2 has been selected for evaluation in the current NTHI MCAT-008 study. The current study will evaluate the impact of a 3rd dose (following a 0-2 month vaccination schedule), either given at 6 months or at 12 months after the first dose. The primary aim is to assess the safety of the additional dose. The study will also investigate how the two schedules improve the persistence of antibody response.

To this end, adults aged 40 to 80 years with a smoking history of at least 10 pack-years, will receive 2 doses of the NTHi-Mcat investigational vaccine at 0 and 2 months in both study arms. Following these 2 doses, one study arm will receive a 3rd dose of the investigational NTHi-Mcat vaccine at 6 months and a placebo control at 12 months (Schedule 1) and the other study arm will receive a placebo control at 6 months and a 3rd dose of the investigational NTHi-Mcat vaccine at 12 months (Schedule 2).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performing any study specific procedure.
* A male or female between, and including, 40 and 80 years of age at the time of the first vaccination.
* Current or former smoker with a cigarette smoking history of ≥ 10 pack-years.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines during the period starting 30 days before the first dose of study vaccines (Day -29 to Day 1), or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the first vaccine dose. For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first and ending 30 days after the last dose of vaccine administration, with the exception of any influenza or pneumococcal vaccine which may be administered ≥ 15 days preceding or following any study vaccine dose.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Previous vaccination with any vaccine containing NTHi and/or Mcat antigens.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of or current autoimmune disease.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥37.5°C. The preferred location for measuring temperature in this study will be the oral cavity or the axilla.
  * Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the first dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Current alcoholism and/or drug abuse.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Diagnosed with a respiratory disorder.
* Has significant disease, in the opinion of the investigator, likely to interfere with the study and/or likely to cause death within the study duration.
* Malignancies within previous 5 years or lymphoproliferative disorders.
* Any other condition that the investigator judges may interfere with study findings.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-09-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- Canada (2):
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Sherbrooke, Quebec
- Germany (2):
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Goch, North Rhine-Westphalia
- United Kingdom (4):
  - GSK Investigational Site, Chesterfield, Derbyshire
  - GSK Investigational Site, Wellingborough, Northamptonshire
  - GSK Investigational Site, Axbridge, Somerset
  - GSK Investigational Site, Chippenham

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Galgani I, Annaratone M, Casula D, Di Maro G, Janssens M, Tasciotti A, Schwarz T, Ferguson M, Arora AK. Safety and immunogenicity of three doses of non-typeable Haemophilus influenzae-Moraxella catarrhalis (NTHi-Mcat) vaccine when administered according to two different schedules: a phase 2, randomised, observer-blind study. Respir Res. 2022 May 4;23(1):114. doi: 10.1186/s12931-022-02019-4. PMID 35509077

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Started | 100 | 100
Completed | 88 | 89
Not Completed | 12 | 11
Not completed — Adverse Event | 2 | 3
Not completed — CONSENT WITHDRAWAL NOT DUE TO ADV. EVENT | 6 | 2
Not completed — Other | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (10.3) | 59.8 (10.1) | 59.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 43 | 89
  Male | 54 | 57 | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 1 | 1
  WHITE | 100 | 99 | 199

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reported With Each Solicited Local Adverse Event (AE) (Any and Grade 3) Within Each Vaccination Schedule
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) injection site.
Time Frame: During the 7-day follow-up period (the day of vaccination + 6 days) after each vaccination administered at Day 1, Day 61, Day 181 and Day 361
Population: Analysis was performed on the Exposed Set (ES) which included all eligible subjects, enrolled in this study, who provided informed consent, had at least one vaccine dose administered and who provided solicited safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 100 | 100
Participants
  Pain, Any, Dose 1 | 64 | 64
  Pain, Grade 3, Dose 1 | 2 | 1
  Pain, Any, Dose 2: number analyzed (Participants) | 92 | 97
  Pain, Any, Dose 2 | 72 | 69
  Pain, Grade 3, Dose 2: number analyzed (Participants) | 92 | 97
  Pain, Grade 3, Dose 2 | 13 | 3
  Pain, Any, Dose 3: number analyzed (Participants) | 89 | 97
  Pain, Any, Dose 3 | 67 | 4
  Pain, Grade 3, Dose 3: number analyzed (Participants) | 89 | 97
  Pain, Grade 3, Dose 3 | 12 | 0
  Pain, Any, Dose 4: number analyzed (Participants) | 84 | 93
  Pain, Any, Dose 4 | 9 | 73
  Pain, Grade 3, Dose 4: number analyzed (Participants) | 84 | 93
  Pain, Grade 3, Dose 4 | 0 | 8
  Redness, Any, Dose 1 | 9 | 18
  Redness, Grade 3, Dose 1 | 0 | 0
  Redness, Any, Dose 2: number analyzed (Participants) | 92 | 97
  Redness, Any, Dose 2 | 12 | 11
  Redness, Grade 3, Dose 2: number analyzed (Participants) | 92 | 97
  Redness, Grade 3, Dose 2 | 0 | 0
  Redness, Any, Dose 3: number analyzed (Participants) | 89 | 97
  Redness, Any, Dose 3 | 13 | 0
  Redness, Grade 3, Dose 3: number analyzed (Participants) | 89 | 97
  Redness, Grade 3, Dose 3 | 1 | 0
  Redness, Any, Dose 4: number analyzed (Participants) | 84 | 93
  Redness, Any, Dose 4 | 1 | 12
  Redness, Grade 3, Dose 4: number analyzed (Participants) | 84 | 93
  Redness, Grade 3, Dose 4 | 0 | 1
  Swelling, Any, Dose 1 | 8 | 10
  Swelling, Grade 3, Dose 1 | 0 | 0
  Swelling, Any, Dose 2: number analyzed (Participants) | 92 | 97
  Swelling, Any, Dose 2 | 7 | 7
  Swelling, Grade 3, Dose 2: number analyzed (Participants) | 92 | 97
  Swelling, Grade 3, Dose 2 | 0 | 0
  Swelling, Any, Dose 3: number analyzed (Participants) | 89 | 97
  Swelling, Any, Dose 3 | 9 | 0
  Swelling, Grade 3, Dose 3: number analyzed (Participants) | 89 | 97
  Swelling, Grade 3, Dose 3 | 1 | 0
  Swelling, Any, Dose 4: number analyzed (Participants) | 84 | 93
  Swelling, Any, Dose 4 | 1 | 10
  Swelling, Grade 3, Dose 4: number analyzed (Participants) | 84 | 93
  Swelling, Grade 3, Dose 4 | 0 | 1

2. Primary Outcome: Number of Subjects Reported With Each Solicited General Adverse Event (AE) (Any and Grade 3) Within Each Vaccination Schedule
Description: Assessed solicited general symptoms were chills, gastrointestinal symptoms (including nausea, vomiting, diarrhoea and/or abdominal pain), fatigue, myalgia, headache and fever [defined Oral cavity or axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.0 °C.
Time Frame: as for outcome 1
Population: Analysis was performed on the Exposed Set which included all eligible subjects, enrolled in this study, who provided informed consent, had at least one vaccine dose administered and who provided solicited safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 100 | 100
Participants
  Chills, Any, Dose 1 | 6 | 5
  Chills, Grade 3, Dose 1 | 0 | 0
  Chills, Any, Dose 2: number analyzed (Participants) | 92 | 97
  Chills, Any, Dose 2 | 13 | 8
  Chills, Grade 3, Dose 2: number analyzed (Participants) | 92 | 97
  Chills, Grade 3, Dose 2 | 4 | 1
  Chills, Any, Dose 3: number analyzed (Participants) | 89 | 97
  Chills, Any, Dose 3 | 12 | 2
  Chills, Grade 3, Dose 3: number analyzed (Participants) | 89 | 97
  Chills, Grade 3, Dose 3 | 4 | 0
  Chills, Any, Dose 4: number analyzed (Participants) | 84 | 93
  Chills, Any, Dose 4 | 2 | 18
  Chills, Grade 3, Dose 4: number analyzed (Participants) | 84 | 93
  Chills, Grade 3, Dose 4 | 1 | 1
  Gastrointestinal symptoms, Any, Dose 1 | 11 | 7
  Gastrointestinal symptoms, Grade 3, Dose 1 | 0 | 0
  Gastrointestinal symptoms, Any, Dose 2: number analyzed (Participants) | 92 | 97
  Gastrointestinal symptoms, Any, Dose 2 | 11 | 10
  Gastrointestinal symptoms, Grade 3, Dose 2: number analyzed (Participants) | 92 | 97
  Gastrointestinal symptoms, Grade 3, Dose 2 | 1 | 1
  Gastrointestinal symptoms, Any, Dose 3: number analyzed (Participants) | 89 | 97
  Gastrointestinal symptoms, Any, Dose 3 | 9 | 7
  Gastrointestinal symptoms, Grade 3, Dose 3: number analyzed (Participants) | 89 | 97
  Gastrointestinal symptoms, Grade 3, Dose 3 | 0 | 0
  Gastrointestinal symptoms, Any, Dose 4: number analyzed (Participants) | 84 | 93
  Gastrointestinal symptoms, Any, Dose 4 | 3 | 15
  Gastrointestinal symptoms, Grade 3, Dose 4: number analyzed (Participants) | 84 | 93
  Gastrointestinal symptoms, Grade 3, Dose 4 | 1 | 1
  Fatigue, Any, Dose 1 | 22 | 16
  Fatigue, Grade 3, Dose 1 | 0 | 1
  Fatigue, Any, Dose 2: number analyzed (Participants) | 92 | 97
  Fatigue, Any, Dose 2 | 28 | 32
  Fatigue, Grade 3, Dose 2: number analyzed (Participants) | 92 | 97
  Fatigue, Grade 3, Dose 2 | 9 | 1
  Fatigue, Any, Dose 3: number analyzed (Participants) | 89 | 97
  Fatigue, Any, Dose 3 | 20 | 13
  Fatigue, Grade 3, Dose 3: number analyzed (Participants) | 89 | 97
  Fatigue, Grade 3, Dose 3 | 4 | 0
  Fatigue, Any, Dose 4: number analyzed (Participants) | 84 | 93
  Fatigue, Any, Dose 4 | 8 | 35
  Fatigue, Grade 3, Dose 4: number analyzed (Participants) | 84 | 93
  Fatigue, Grade 3, Dose 4 | 3 | 5
  Myalgia, Any, Dose 1 | 17 | 16
  Myalgia, Grade 3, Dose 1 | 1 | 0
  Myalgia, Any, Dose 2: number analyzed (Participants) | 92 | 97
  Myalgia, Any, Dose 2 | 22 | 23
  Myalgia, Grade 3, Dose 2: number analyzed (Participants) | 92 | 97
  Myalgia, Grade 3, Dose 2 | 7 | 1
  Myalgia, Any, Dose 3: number analyzed (Participants) | 89 | 97
  Myalgia, Any, Dose 3 | 20 | 3
  Myalgia, Grade 3, Dose 3: number analyzed (Participants) | 89 | 97
  Myalgia, Grade 3, Dose 3 | 6 | 0
  Myalgia, Any, Dose 4: number analyzed (Participants) | 84 | 93
  Myalgia, Any, Dose 4 | 4 | 28
  Myalgia, Grade 3, Dose 4: number analyzed (Participants) | 84 | 93
  Myalgia, Grade 3, Dose 4 | 1 | 5
  Headache, Any, Dose 1 | 13 | 15
  Headache, Grade 3, Dose 1 | 0 | 1
  Headache, Any, Dose 2: number analyzed (Participants) | 92 | 97
  Headache, Any, Dose 2 | 24 | 21
  Headache, Grade 3, Dose 2: number analyzed (Participants) | 92 | 97
  Headache, Grade 3, Dose 2 | 2 | 1
  Headache, Any, Dose 3: number analyzed (Participants) | 89 | 97
  Headache, Any, Dose 3 | 24 | 7
  Headache, Grade 3, Dose 3: number analyzed (Participants) | 89 | 97
  Headache, Grade 3, Dose 3 | 4 | 0
  Headache, Any, Dose 4: number analyzed (Participants) | 84 | 93
  Headache, Any, Dose 4 | 5 | 27
  Headache, Grade 3, Dose 4: number analyzed (Participants) | 84 | 93
  Headache, Grade 3, Dose 4 | 1 | 1
  Fever, Any, Dose 1 | 3 | 3
  Fever, Grade 3, Dose 1 | 0 | 0
  Fever, Any, Dose 2: number analyzed (Participants) | 92 | 97
  Fever, Any, Dose 2 | 3 | 6
  Fever, Grade 3, Dose 2: number analyzed (Participants) | 92 | 97
  Fever, Grade 3, Dose 2 | 0 | 0
  Fever, Any, Dose 3: number analyzed (Participants) | 89 | 97
  Fever, Any, Dose 3 | 4 | 2
  Fever, Grade 3, Dose 3: number analyzed (Participants) | 89 | 97
  Fever, Grade 3, Dose 3 | 0 | 0
  Fever, Any, Dose 4: number analyzed (Participants) | 84 | 93
  Fever, Any, Dose 4 | 3 | 5
  Fever, Grade 3, Dose 4: number analyzed (Participants) | 84 | 93
  Fever, Grade 3, Dose 4 | 0 | 0

3. Primary Outcome: Number of Subjects Reported With Any Unsolicited Adverse Event (AE) Within Each Vaccination Schedule
Description: An AE is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: During the 30-day follow-up period (the day of vaccination + 29 days) after each vaccination administered at Day 1, Day 61, Day 181 and Day 361
Population: Analysis was performed on the Exposed Set which included all eligible subjects, enrolled in this study, who provided informed consent, had at least one vaccine dose administered and who provided unsolicited safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 100 | 100
Participants
  Dose 1 | 16 | 20
  Dose 2: number analyzed (Participants) | 93 | 98
  Dose 2 | 15 | 20
  Dose 3: number analyzed (Participants) | 90 | 97
  Dose 3 | 13 | 11
  Dose 4: number analyzed (Participants) | 85 | 93
  Dose 4 | 7 | 9

4. Primary Outcome: Number of Subjects Reported With Any Serious Adverse Event (SAE) Within Each Vaccination Schedule
Description: An SAE is defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity in a subject or was a congenital anomaly/birth defect in the offspring of a study subject. AE(s) considered as SAE(s) also include invasive or malignant cancers, intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalization, as per the medical or scientific judgement of the physician.
Time Frame: From first vaccination (Day 1) up to Day 541 (an average of 18 months)
Population: Analysis was performed on the Exposed set which included all eligible subjects, enrolled in this study, who provided informed consent, had at least one vaccine dose administered and who provided safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 100 | 100
Participants | 12 | 8

5. Primary Outcome: Number of Subjects Reported With Any Potential Immune-mediated Diseases (pIMDs) Within Each Vaccination Schedule
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From first vaccination (Day 1) up to Day 541 (an average of 18 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 100 | 100
Participants | 3 | 3

6. Secondary Outcome: Number of Subjects Reported With Any SAE Within Each Vaccination Schedule
Description: as for outcome 4
Time Frame: From Day 541 up to Day 721 (an average of 6 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 100 | 100
Participants | 0 | 2

7. Secondary Outcome: Number of Subjects Reported With Any pIMDs Within Each Vaccination Schedule
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From Day 541 up to Day 721 (an average of 6 months)
Population: Analysis was performed on the Exposed set which included all eligible subjects, enrolled in this study, who provided informed consent, had at least one vaccine dose.
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 100 | 100
Participants | 0 | 0

8. Secondary Outcome: Anti-Protein D (PD) Antibody Concentrations, as Measured by ELISA, Within Each Vaccination Schedule
Description: Anti-Protein D (PD) antibody concentrations as determined by Enzyme-linked Immunosorbent Assay (ELISA), and expressed as geometric mean concentrations (GMCs) in ELISA unit per milliliter (EU/mL). Calculation of the GMCs are performed by taking the anti-logarithm in base 10 (anti-log10) of the mean of the log10 concentration transformations. Antibody concentrations below the assay cut-off (153 EU/mL) is given an arbitrary value of half the assay cut-off for the purpose of GMC calculation.
Time Frame: At Day 1, Day 91, Day 181, Day 211, Day 361, Day 391, Day 541 and Day 721
Population: Analysis was performed on the Per Protocol Set which included all eligible subjects enrolled in this study, who provided informed consent, who complied with the vaccination schedule and who provided immunogenicity data according to blood sample timings specified in the protocol
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 82 | 87
EU/mL
  Day 1 | 88 [79.2 to 97.9] | 88.1 [79.8 to 97.2]
  Day 91: number analyzed (Participants) | 79 | 82
  Day 91 | 1365.5 [1073.0 to 1737.8] | 1394.1 [1116.9 to 1740.1]
  Day 181: number analyzed (Participants) | 81 | 87
  Day 181 | 853.4 [665.4 to 1094.6] | 835.6 [665.4 to 1049.3]
  Day 211: number analyzed (Participants) | 81 | 84
  Day 211 | 2338 [1840.1 to 2970.8] | 679 [541.7 to 850.9]
  Day 361 | 1199 [942.8 to 1524.9] | 483.1 [386.4 to 603.9]
  Day 391: number analyzed (Participants) | 81 | 82
  Day 391 | 1064.1 [829.4 to 1365.2] | 2677 [2111.4 to 3394.1]
  Day 541: number analyzed (Participants) | 80 | 84
  Day 541 | 826.5 [646.3 to 1057.0] | 1346.4 [1072.1 to 1690.8]
  Day 721: number analyzed (Participants) | 77 | 79
  Day 721 | 679.6 [529.5 to 872.1] | 900.4 [716.1 to 1132.2]

9. Secondary Outcome: Anti-Protein E (PE) Antibody Concentrations, as Measured by ELISA, Within Each Vaccination Schedule
Description: Anti-Protein E (PE) antibody concentrations as determined by ELISA, and expressed in EU/mL. Calculation of the GMCs are performed by taking the anti-logarithm in base 10 (anti-log10) of the mean of the log10 concentration transformations. Antibody concentrations below the assay cut-off (16 EU/mL) is given an arbitrary value of half the assay cut-off for the purpose of GMC calculation.
Time Frame: At Day 1, Day 91, Day 181, Day 211, Day 361, Day 391, Day 541 and Day 721
Population: Analysis was performed on the Per Protocol Set which included all eligible subjects, enrolled in this study, who provided informed consent, who complied with the vaccination schedule and who provided immunogenicity data according to blood sample timings specified in the protocol
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 82 | 87
EU/mL
  Day 1 | 19.6 [15.1 to 25.5] | 18.4 [14.5 to 23.5]
  Day 91: number analyzed (Participants) | 79 | 82
  Day 91 | 5867.9 [4644.4 to 7413.8] | 5896.7 [4755.2 to 7312.3]
  Day 181: number analyzed (Participants) | 81 | 87
  Day 181 | 2649.1 [2113.3 to 3320.7] | 2787.1 [2266.0 to 3428.0]
  Day 211: number analyzed (Participants) | 80 | 84
  Day 211 | 7557.1 [6107.9 to 9350.0] | 2309.9 [1892.1 to 2819.8]
  Day 361 | 2735.3 [2196.7 to 3406.1] | 1298 [1058.6 to 1591.6]
  Day 391: number analyzed (Participants) | 81 | 82
  Day 391 | 2604.2 [2118.3 to 3201.5] | 9339.4 [7670.2 to 11372.0]
  Day 541: number analyzed (Participants) | 80 | 84
  Day 541 | 1762.2 [1443.9 to 2150.6] | 3620.7 [3009.9 to 4355.4]
  Day 721: number analyzed (Participants) | 77 | 79
  Day 721 | 1348.3 [1085.6 to 1674.7] | 1942.0 [1591.0 to 2370.5]

10. Secondary Outcome: Anti-Type IV Pili Subunit (PilA) Antibody Concentrations, as Measured by ELISA, Within Each Vaccination Schedule
Description: Anti-type IV pili subunit (PilA) antibody concentrations as determined by ELISA, and expressed in EU/mL. Calculation of the GMCs are performed by taking the anti-logarithm in base 10 (anti-log10) of the mean of the log10 concentration transformations. Antibody concentrations below the assay cut-off (8 EU/mL) is given an arbitrary value of half the assay cut-off for the purpose of GMC calculation.
Time Frame: At Day 1, Day 91, Day 181, Day 211, Day 361, Day 391, Day 541 and Day 721
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 82 | 87
EU/mL
  Day 1 | 10.9 [8.5 to 14.2] | 8.3 [6.5 to 10.5]
  Day 91: number analyzed (Participants) | 79 | 82
  Day 91 | 992.5 [747.2 to 1318.5] | 893.1 [688.6 to 1158.3]
  Day 181: number analyzed (Participants) | 81 | 87
  Day 181 | 589.3 [442.8 to 784.3] | 504.2 [388.4 to 654.3]
  Day 211: number analyzed (Participants) | 81 | 84
  Day 211 | 1191.7 [920.0 to 1543.6] | 396.3 [310.9 to 505.2]
  Day 361 | 546.6 [418.1 to 714.5] | 250.3 [195.3 to 320.7]
  Day 391: number analyzed (Participants) | 81 | 82
  Day 391 | 456.4 [360.7 to 577.6] | 1163.9 [931.1 to 1454.9]
  Day 541: number analyzed (Participants) | 80 | 84
  Day 541 | 330.4 [260.5 to 419.1] | 524.3 [421.0 to 653.1]
  Day 721: number analyzed (Participants) | 77 | 79
  Day 721 | 242.9 [186.4 to 316.5] | 305.5 [239.8 to 389.2]

11. Secondary Outcome: Anti-Ubiquitous Surface Protein A2 of Moraxella Catarrhalis (UspA2) Antibody Concentrations, as Measured by ELISA, Within Each Vaccination Schedule
Description: Anti-ubiquitous surface protein A2 of Moraxella catarrhalis (UspA2) antibody concentrations as determined by ELISA, and expressed in EU/mL. Calculation of the GMCs are performed by taking the anti-logarithm in base 10 (anti-log10) of the mean of the log10 concentration transformations. Antibody concentrations below the assay cut-off (28 EU/mL) is given an arbitrary value of half the assay cut-off for the purpose of GMC calculation.
Time Frame: At Day 1, Day 91, Day 181, Day 211, Day 361, Day 391, Day 541 and Day 721
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 82 | 87
EU/mL
  Day 1 | 682.4 [544.4 to 855.4] | 544.9 [441.8 to 672.1]
  Day 91: number analyzed (Participants) | 79 | 82
  Day 91 | 1364.5 [1217.6 to 1529.1] | 1159.7 [1044.8 to 1287.2]
  Day 181: number analyzed (Participants) | 81 | 87
  Day 181 | 1019.7 [920.9 to 1129.0] | 915.2 [834.1 to 1004.3]
  Day 211: number analyzed (Participants) | 81 | 84
  Day 211 | 1270.9 [1138.1 to 1419.2] | 864.6 [779.5 to 959.1]
  Day 361 | 885.8 [801.7 to 978.8] | 730 [665.6 to 800.6]
  Day 391: number analyzed (Participants) | 81 | 82
  Day 391 | 909.9 [818.5 to 1011.4] | 1142.8 [1033.9 to 1263.3]
  Day 541: number analyzed (Participants) | 80 | 84
  Day 541 | 898.2 [811.5 to 994.2] | 847.4 [771.6 to 930.7]
  Day 721: number analyzed (Participants) | 77 | 79
  Day 721 | 790.6 [705.1 to 886.6] | 715.2 [644.0 to 794.1]

12. Secondary Outcome: Number of Seropositive Subjects for Anti-PD Antibody, as Measured by ELISA, Within Each Vaccination Schedule
Description: A Seropositive subject is defined as a subject whose antibody concentration is greater than or equal to the assay cut off (i.e. the ELISA lower limit of quantification = 153 EU/mL).Antibody concentrations as determined by Enzyme-linked Immunosorbent Assay (ELISA), and expressed in EU/mL.
Time Frame: At Day 1, Day 91, Day 181, Day 211, Day 361, Day 391, Day 541 and Day 721
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 82 | 87
Participants
  Day 1 | 7 | 12
  Day 91: number analyzed (Participants) | 79 | 82
  Day 91 | 78 | 80
  Day 181: number analyzed (Participants) | 81 | 87
  Day 181 | 75 | 80
  Day 211: number analyzed (Participants) | 81 | 84
  Day 211 | 81 | 75
  Day 361 | 78 | 71
  Day 391: number analyzed (Participants) | 81 | 82
  Day 391 | 77 | 81
  Day 541: number analyzed (Participants) | 80 | 84
  Day 541 | 76 | 79
  Day 721: number analyzed (Participants) | 77 | 79
  Day 721 | 72 | 74

13. Secondary Outcome: Number of Seropositive Subjects for Anti-PE Antibody, as Measured by ELISA, Within Each Vaccination Schedule
Description: A Seropositive subject is defined as a subject whose antibody concentration is greater than or equal to the assay cut off (i.e. the ELISA lower limit of quantification = 16 EU/mL). Antibody concentrations as determined by Enzyme-linked Immunosorbent Assay (ELISA), and expressed in EU/mL.
Time Frame: At Day 1, Day 91, Day 181, Day 211, Day 361, Day 391, Day 541 and Day 721
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 82 | 87
Participants
  Day 1 | 43 | 43
  Day 91: number analyzed (Participants) | 79 | 82
  Day 91 | 79 | 82
  Day 181: number analyzed (Participants) | 81 | 87
  Day 181 | 81 | 87
  Day 211: number analyzed (Participants) | 80 | 84
  Day 211 | 80 | 84
  Day 361 | 82 | 87
  Day 391: number analyzed (Participants) | 81 | 82
  Day 391 | 81 | 82
  Day 541: number analyzed (Participants) | 80 | 84
  Day 541 | 80 | 84
  Day 721: number analyzed (Participants) | 77 | 79
  Day 721 | 77 | 79

14. Secondary Outcome: Number of Seropositive Subjects for Anti- PilA Antibody, as Measured by ELISA, Within Each Vaccination Schedule
Description: A Seropositive subject is defined as a subject whose antibody concentration is greater than or equal to the assay cut off (i.e. the ELISA lower limit of quantification = 8 EU/mL).Antibody concentrations as determined by Enzyme-linked Immunosorbent Assay (ELISA), and expressed in EU/mL.
Time Frame: At Day 1, Day 91, Day 181, Day 211, Day 361, Day 391, Day 541 and Day 721
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 82 | 87
Participants
  Day 1 | 40 | 36
  Day 91: number analyzed (Participants) | 79 | 82
  Day 91 | 79 | 82
  Day 181: number analyzed (Participants) | 81 | 87
  Day 181 | 81 | 87
  Day 211: number analyzed (Participants) | 81 | 84
  Day 211 | 81 | 83
  Day 361 | 82 | 84
  Day 391: number analyzed (Participants) | 81 | 82
  Day 391 | 81 | 82
  Day 541: number analyzed (Participants) | 80 | 84
  Day 541 | 80 | 84
  Day 721: number analyzed (Participants) | 77 | 79
  Day 721 | 75 | 79

15. Secondary Outcome: Number of Seropositive Subjects for Anti- UspA2 Antibody, as Measured by ELISA, Within Each Vaccination Schedule
Description: A Seropositive subject is defined as a subject whose antibody concentration is greater than or equal to the assay cut off (i.e. the ELISA lower limit of quantification = 28 EU/mL).Antibody concentrations as determined by Enzyme-linked Immunosorbent Assay (ELISA), and expressed in EU/mL.
Time Frame: At Day 1, Day 91, Day 181, Day 211, Day 361, Day 391, Day 541 and Day 721
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 82 | 87
Participants
  Day 1 | 82 | 87
  Day 91: number analyzed (Participants) | 79 | 82
  Day 91 | 79 | 82
  Day 181: number analyzed (Participants) | 81 | 87
  Day 181 | 81 | 87
  Day 211: number analyzed (Participants) | 81 | 84
  Day 211 | 81 | 84
  Day 361 | 82 | 87
  Day 391: number analyzed (Participants) | 81 | 82
  Day 391 | 81 | 82
  Day 541: number analyzed (Participants) | 80 | 84
  Day 541 | 80 | 84
  Day 721: number analyzed (Participants) | 77 | 79
  Day 721 | 77 | 79

16. Secondary Outcome: Frequency of Specific Cluster of Differentiation 4 (CD4+) T-cells Producing 2 or More Markers Upon in Vitro Stimulation With the Antigen, by NTHi and Mcat Antigens
Description: Frequency of specific CD4+ T-cells were measured by flow cytometry intracellular cytokine staining (ICS) expressing two or more markers [such as Interleukin-2 (IL-2), IL-13, IL-17, Interferon-γ (IFN-γ), Tumor Necrosis Factor-α (TNF-α) and Cluster of Differentiation 40 Ligand (CD40L)]. The frequency of specific CD4+ T-cells are summarized with following descriptive statistics: Mean and standard deviation (SD) against each antigen (PD, PE,PilA and UspA2), by group and at each time point for which blood samples were collected for Cell-Mediated Immunity (CMI). The CMI sub-cohort subjects were selected from sites able to process the blood samples according to GSK procedures for peripheral blood mononuclear cell (PBMC) preparation.
Time Frame: At Day 1, Day 91, Day 181, Day 211, Day 361 and Day 391
Population: Analysis was performed on a subset of subjects (CMI sub cohort), which included approximately 20 subjects in each group,for which additional blood sample was taken at each pre-defined timepoint.
Measure: Mean (Standard Deviation); unit: CD4+ T-cells/million cells
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
Number analyzed (Participants) | 21 | 19
CD4+ T-cells/million cells
  NTHi.PD, Day 1 | 76.995 (142.760) | 55.173 (109.539)
  NTHi.PD, Day 91: number analyzed (Participants) | 19 | 19
  NTHi.PD, Day 91 | 865.933 (919.585) | 1076.136 (970.670)
  NTHi.PD, Day 181: number analyzed (Participants) | 17 | 19
  NTHi.PD, Day 181 | 381.265 (356.496) | 463.939 (558.441)
  NTHi.PD, Day 211: number analyzed (Participants) | 17 | 19
  NTHi.PD, Day 211 | 664.044 (610.930) | 518.104 (513.462)
  NTHi.PD, Day 361: number analyzed (Participants) | 17 | 17
  NTHi.PD, Day 361 | 444.129 (520.204) | 378.78 (456.970)
  NTHi.PD, Day 391: number analyzed (Participants) | 17 | 17
  NTHi.PD, Day 391 | 321.28 (316.073) | 761.605 (974.791)
  NTHi.PE, Day 1 | 28.869 (44.944) | 21.223 (38.682)
  NTHi.PE, Day 91: number analyzed (Participants) | 19 | 19
  NTHi.PE, Day 91 | 1406.663 (1900.558) | 926.809 (785.046)
  NTHi.PE, Day 181: number analyzed (Participants) | 17 | 19
  NTHi.PE, Day 181 | 551.444 (635.058) | 352.471 (403.081)
  NTHi.PE, Day 211: number analyzed (Participants) | 17 | 19
  NTHi.PE, Day 211 | 986.138 (1570.491) | 463.076 (395.158)
  NTHi.PE, Day 361: number analyzed (Participants) | 17 | 17
  NTHi.PE, Day 361 | 636.539 (995.486) | 305.772 (337.400)
  NTHi.PE, Day 391: number analyzed (Participants) | 17 | 17
  NTHi.PE, Day 391 | 590.426 (714.051) | 481.133 (533.658)
  NTHi.PilA, Day 1 | 81.03 (178.861) | 79.205 (210.642)
  NTHi.PilA, Day 91: number analyzed (Participants) | 19 | 19
  NTHi.PilA, Day 91 | 615.698 (686.114) | 523.195 (493.956)
  NTHi.PilA, Day 181: number analyzed (Participants) | 17 | 19
  NTHi.PilA, Day 181 | 356.275 (350.909) | 265.097 (267.351)
  NTHi.PilA, Day 211: number analyzed (Participants) | 17 | 19
  NTHi.PilA, Day 211 | 524.754 (654.443) | 257.806 (252.382)
  NTHi.PilA, Day 361: number analyzed (Participants) | 17 | 17
  NTHi.PilA, Day 361 | 341.58 (433.970) | 205.388 (220.979)
  NTHi.PilA, Day 391: number analyzed (Participants) | 17 | 17
  NTHi.PilA, Day 391 | 334.088 (300.114) | 368.693 (354.449)
  M catarrhalis.UspA2, Day 1 | 85.785 (99.051) | 53.391 (80.742)
  M catarrhalis.UspA2, Day 91: number analyzed (Participants) | 19 | 19
  M catarrhalis.UspA2, Day 91 | 964.521 (709.134) | 730.725 (575.778)
  M catarrhalis.UspA2, Day 181: number analyzed (Participants) | 17 | 19
  M catarrhalis.UspA2, Day 181 | 559.062 (524.096) | 355.992 (346.277)
  M catarrhalis.UspA2, Day 211: number analyzed (Participants) | 17 | 19
  M catarrhalis.UspA2, Day 211 | 846.177 (750.349) | 424.981 (329.334)
  M catarrhalis.UspA2, Day 361: number analyzed (Participants) | 17 | 17
  M catarrhalis.UspA2, Day 361 | 635.022 (617.485) | 347.65 (363.499)
  M catarrhalis.UspA2, Day 391: number analyzed (Participants) | 17 | 17
  M catarrhalis.UspA2, Day 391 | 545.436 (464.272) | 474.238 (446.236)

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected during the 7-day follow-up (FU) period after any vaccination. Unsolicited AEs during the 30-day follow-up (FU) period after any vaccination and SAEs from Day 1 to Day 721
Arm/Group | Schedule 0-2-6 Group | Schedule 0-2-12 Group
All-Cause Mortality (participants affected / at risk) | 1/100 | 2/100
Serious Adverse Events (participants affected / at risk) | 12/100 | 9/100
Other Adverse Events (participants affected / at risk) | 93/100 | 97/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Schedule 0-2-6 Group (N=100) | Schedule 0-2-12 Group (N=100)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Right ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (3)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tooth injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Cerebral artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Conversion disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Schedule 0-2-6 Group (N=100) | Schedule 0-2-12 Group (N=100)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 25 (34) | 28 (40)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Administration site pruritus (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Chills (General disorders) | 24 (33) | 25 (34)
Fatigue (General disorders) | 44 (79) | 50 (97)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 2 (2) | 2 (2)
Injection site erythema (General disorders) | 21 (35) | 28 (41)
Injection site pain (General disorders) | 89 (213) | 92 (210)
Injection site pruritus (General disorders) | 0 (0) | 1 (1)
Injection site swelling (General disorders) | 16 (25) | 20 (27)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 11 (13) | 13 (16)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0)
Alveolar osteitis (Infections and infestations) | 1 (2) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Gingival abscess (Infections and infestations) | 0 (0) | 1 (1)
Infected bite (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (6) | 6 (6)
Ophthalmic herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Weight increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 38 (63) | 41 (73)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 39 (69) | 41 (71)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 4 (4)
Illness (General disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/27/NCT03443427/Prot_001.pdf
  • Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT03443427/SAP_000.pdf